CLINICAL TRIAL: NCT04618094
Title: Feasibility and Acceptance of High Intensity Interval Training in the Prehabilitation of Patients Suffering From Gynecological Cancers - a Randomized Controlled Pilot Study
Brief Title: Prehabilitation in Patients Suffering From Gynecological Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefano Palma, Principal Investigator, PhD student, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Prehab
Record Dates: First submitted 2020-10-15; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Prehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval group (Experimental)
  Interventions: Other: bicycle ergometer training with different intensities
- Moderate continous intensity group (Active Comparator)
  Interventions: Other: bicycle ergometer training with different intensities
- non-exercising group (No Intervention)

INTERVENTIONS:
Other: bicycle ergometer training with different intensities — Following a 10-min warm-up phase at a constant work load below ventilatory threshold, participants of the high intensity interval group perform repeated high intensity exercise bouts, followed by an active recovery on a bicycle ergometer. The comparative group perform a constant moderate intensity with the same mean workload. The cool-down phase is 5 min with a constant work load for both groups.
  Arms: High intensity interval group; Moderate continous intensity group

SUMMARY:
In 2016, 2216 Austrian women (= 10% of all new cancer cases) were diagnosed with gynecological tumors. Depending on stage and entity, a main primary therapy option is the surgical tumor resection. In the phase of Prehabilitation (= the time frame from diagnosis to surgical intervention) supportive therapy options such as individualized exercise interventions potentially improve recovery and postoperative outcomes after surgical interventions. The primary aim of this study is to investigate the feasibility and acceptance of a prehabilitation training intervention with high-intensity interval training compared to a conventional moderate intensity continuous training and a non-training collective. Secondary goals are the investigation of the effectiveness of threshold-based intensity prescriptions and the impact on quality of life, fatigue, anxiety, depression, sexuality and ability to work.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically verified cervical carcinoma (ICD10-C53) or
* endometrial carcinoma (ICD10-C54) or
* ovarian carcinoma (ICD10-C56)
* planned primary/adjuvant surgery or medical training therapy
* oncological release for medical training therapy
* Eastern cooperative oncology group performance status (ECOG) 0-II
* Age >18a to 80
* mental aptitude to participate in the study

Exclusion Criteria:

* serious orthopaedic, rheumatological, neurological, oncological and cardiovascular diseases which are incompatible with a training intervention
* general contraindications for exercise ergometry according to the guidelines of the austrian society of cardiology
* osseous or cerebral metastasis
* participation in a training study in the last year or already before cancer diagnosis with high training volumes (>150min moderate / >75min more intensive endurance training per week)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
adherence to the exercise intervention | 4 to 8 weeks
  rate of completed exercise sessions as a measure of feasibility and acceptance

SECONDARY OUTCOMES:
cardiovascular fitness | 4 to 8 Weeks
  determined by VO2max
workability | 4 to 8 weeks
  determined by the workability index questionnaire; minimum value 7, maximum value 49, higher values indicating better results
Health related Quality of life: questionnaire | 4 to 8 weeks
  determined by the European Organisation for Research and Treatment of Cancer Quality of Life questionnaire, minimum value 30, maximum value 126, higher scores indicating higher quality of life
Anxiety and depression | 4 to 8 weeks
  determined by the Hospital Anxiety and Depression Scale questionnaire, minimum value 14, maximum value 56, higher values indicating higher depression levels
handgrip strength | 4 to 8 weeks
  determined by the handgrip dynamometer
body composition | 4 to 8 weeks
  determined by bioimpedance analysis
Cholesterol | 4 to 8 weeks
  Laboratory parameter in mg/ml as a part of the evaluation for cardiovascular risk factors
Thyreoglobulin | 4 to 8 weeks
  Laboratory parameter in µg/ml as a part of the evaluation for cardiovascular risk factors
hemoglobin A1c | 4 to 8 weeks
  Laboratory parameter in % as a part of the evaluation for cardiovascular risk factors
Brain natriuretic peptide | 4 to 8 weeks
  Laboratory parameter in pg/ml as a part of the evaluation for cardiovascular risk factors
Troponin T | 4 to 8 weeks
  Laboratory parameter in µg/ml as a part of the evaluation for cardiovascular risk factors
Creatin Kinase | 4 to 8 weeks
  Laboratory parameter in U/l as a part of the evaluation for cardiovascular risk factors
C-reactive protein | 4 to 8 weeks
  Laboratory parameter in mg/l as a part of the evaluation for inflammation
interleukin 1 | 4 to 8 Weeks
  Laboratory parameter in ng/ml as a part of the evaluation for inflammation
interleukin 6 | 4 to 8 weeks
  Laboratory parameter in ng/ml as a part of the evaluation for inflammation
Tumor Necrosis Factor alpha | 4 to 8 weeks
  Laboratory parameter in pg/ml as a part of the evaluation for inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palma, MD, Principal Investigator — Medical University of Vienna, Waehringer Guertel 18-20, 1090 Vienna, Austria

IPD SHARING:
Plan to Share IPD: No